CLINICAL TRIAL: NCT04265898
Title: Validating the Digital Virginia Tech Carilion Cognitive Examination - A Unique Tool for Cognitive Assessment
Brief Title: Validating the Digital Virginia Tech Carilion Cognitive Examination
Acronym: VTC-Cog
Status: Withdrawn | Type: Observational
Why Stopped: The study did not receive IRB approval and was withdrawn by the PI on April 9, 2020.
Sponsor: Carilion Clinic (Other)
Collaborators: Digitally Enhanced Screening Applications (Industry)
Responsible Party: Sponsor
Other Study IDs: VTC-Cog 19-554
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Cognitive Change

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Test Group: Reported mild cognitive deficits
  Interventions: Device: The Digital Virginia Tech Carilion Cognitive Examination
- Control Group: No cognitive deficits
  Interventions: Device: The Digital Virginia Tech Carilion Cognitive Examination

INTERVENTIONS:
Device: The Digital Virginia Tech Carilion Cognitive Examination — Completion of a newly developed digital cognitive screen

SUMMARY:
Currently, cognitive screening is performed in-person after the individual expresses symptoms or it is noticed by someone close to them and are largely done in clinical settings. The digital Virginia Tech Carilion Cognitive Examination (VTC-Cog) utilizes smart devices and allows for the early establishment of an individual's cognitive baseline. VTC-Cog has been designed to test all major aspects of cognition, as currently assessed using the Montreal Cognitive Assessment (MoCA) and Mini-Mental Status Examination (MMSE) but on a digital platform. The VTC-Cog allows for standardized scoring with no clinician bias and provides a clinician report that breaks down distinct changes in different areas of cognition (executive, visuospatial, memory, etc.) in order to refine clinician analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-80 years
* No current diagnosis of dementia
* Current stable mental health
* English speaker
* Carilion Clinic Medical Provider

Exclusion Criteria:

* <50 years old or >80 years old
* Current diagnosis of dementia
* Unstable mental health
* Non-English speaker
* Medical provider outside the Carilion Clinic system

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants must be 50-80 years old with no diagnosis of dementia who speak English, have no acute mental health concerns, and have a Carilion Clinic medical provider.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Validation of the Digital Virginia Tech Carilion Cognitive Examination against the Montreal Cognitive Assessment | 18-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Azziza Bankole, MD, Principal Investigator — Physician